CLINICAL TRIAL: NCT06247436
Title: Alternations in Body Composition of Tonsillectomy Patients During the Recovery Period
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OGYÉI/56432-2/2023
Record Dates: First submitted 2023-10-17; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-10

CONDITIONS: Tonsil Disease
Keywords: body composition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Branch Chained Amino Acids-4mg (Experimental): 4g BCAA, solved in water, twice daily
  Interventions: Dietary Supplement: Branch Chained Amino Acids
- Control (No Intervention): no consumption

INTERVENTIONS:
Dietary Supplement: Branch Chained Amino Acids — postoperative BCAA consumption
  Arms: Branch Chained Amino Acids-4mg

SUMMARY:
The body composition of individuals undergoing tonsillectomy is assessed through bioimpedance-based measurements conducted immediately before the surgery, as well as on the 7th and 21st days during the postoperative period.

DETAILED DESCRIPTION:
In the context of interventions affecting the upper alimentary canal-like tonsillectomy-, it is advisable to adhere to a gentle diet until complete wound healing. Additionally, patients may need to modify their eating habits due to discomfort during swallowing. Physical activity is strictly prohibited during this recovery phase, which poses a risk of muscle loss.

Branched-chain amino acids (BCAAs) play a crucial role in sports nutrition. Unlike other amino acids, BCAAs can be directly utilized by muscles without involving the liver. They serve as an immediate energy source for muscles or contribute to the synthesis of new muscle proteins, helping to prevent muscle loss.

At the same time, the investigators also examined the changes that could be detected in the blood and were possibly related to dietary habits.

ELIGIBILITY:
Inclusion Criteria:

* indication of tonsillectomy
* age between 20-40 years

Exclusion Criteria:

* metabolic diseases,
* haematologic disorders

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
The postoperative changes of body weight (kg) after tonsillectomy | 21 days
  In this study the investigators used Inbody 270, a body bomposition analyzer based on multi-frequency Bioelectrical Impedance Analysis(BIA) method that calculated specific body component by differences in impedance indexes of fat, muscle and extracellular body fluid. Weight alternation was registered in kg.
The postoperative changes of skeletal muscle mass (kg) after tonsillectomy | 21 days
  In this study the investigators used Inbody 270, a body bomposition analyzer based on multi-frequency Bioelectrical Impedance Analysis(BIA) method that calculated specific body component by differences in impedance indexes of fat, muscle and extracellular body fluid. SMM-Skeletal Muscle Mass alteration was registered in kg
The postoperative changes of Body Fat Mass (kg) after tonsillectomy | 21 days
  In this study the investigators used Inbody 270, a body bomposition analyzer based on multi-frequency Bioelectrical Impedance Analysis(BIA) method that calculated specific body component by differences in impedance indexes of fat, muscle and extracellular body fluid. BFM-Body Fat Mass alteration was registered in kg.
The postoperative changes of Body Mass Index (kg/m2) after tonsillectomy | 21 days
  Body weight -registered with InBody 270 - and height of the patient -that not changes in the 3 weeks of time frame of the study- will be combined to report BMI in kg/m2
The postoperative changes of Percent Body Fat (%) after tonsillectomy | 21 days
  In this study the investigators used Inbody 270, a body bomposition analyzer based on multi-frequency Bioelectrical Impedance Analysis(BIA) method that calculated specific body component by differences in impedance indexes of fat, muscle and extracellular body fluid. ), PBF-Percent Body Fat alteration was registered is %
The postoperative changes of Total Body Water (liter) after tonsillectomy | 21 days
  In this study the investigators used Inbody 270, a body bomposition analyzer based on multi-frequency Bioelectrical Impedance Analysis(BIA) method that calculated specific body component by differences in impedance indexes of fat, muscle and extracellular body fluid. TBW-Total Body Water alteration was registered in liter
examination of changes in blood count (mmol/l) | 21 days
  changes in triglyceride, HDL, LDL, Na, K, Ca, Mg, Carbamide, Kreatinine in Units of Measure: mmol/l
determination of changes in blood parametersof Liver Function (U/l) | 21 days
  alterations of GOT,GGT,GPT values in Units of Measure: U/l

SECONDARY OUTCOMES:
effects of branched chain amino acid consumption | 21 days
  determination of the skeletal muscle mass loss in kg after BCAA consumption

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Kiricsi, MD, PhD, Principal Investigator — Szeged University
Locations (1):
- Universitiy of Szeged, Department of Otorhinolaryngology, Head and Neck Surgery, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No